CLINICAL TRIAL: NCT01147003
Title: A 12-week, Multi-center, Randomized, Double-blind, Placebo-controlled Efficacy and Safety Study Examining Seizure Frequency of BGG492 Capsules as Adjunctive Treatment in Patients With Partial Onset Seizures
Brief Title: Efficacy and Safety of BGG492 as Adjunctive Treatment in Patients With Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBGG492A2207; 2009-017961-52 (EudraCT Number)
Record Dates: First submitted 2010-06-15; First posted 2010-06-22 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-03

CONDITIONS: Partial Onset Seizures
Keywords: Seizure frequency; nervous system diseases; brain diseases; neurologic manifestations; adjunctive treatment; AEDs; antiepileptic drug
MeSH Terms: conditions — Nervous System Diseases; Brain Diseases; Neurologic Manifestations | interventions — Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- BGG492 low dose (Experimental)
  Interventions: Drug: Investigational new drug, company code: BGG492
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BGG492 high dose (Experimental)
  Interventions: Drug: Investigational new drug, company code: BGG492

INTERVENTIONS:
Drug: Investigational new drug, company code: BGG492
  Arms: BGG492 low dose
Drug: Placebo
  Arms: Placebo
Drug: Investigational new drug, company code: BGG492
  Arms: BGG492 high dose

SUMMARY:
This study will assess the efficacy and safety of BGG492 as adjunctive treatment in patients with partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥ 50 kg (110 lb) of weight.
* A diagnosis of epilepsy (≥ 2 years prior to screening) with partial seizures with or without secondarily generalized seizures.
* Uncontrolled partial seizures despite having been treated with at least two different antiepileptic drugs (AEDs) within the last 2 years prior to screening.
* At least 4 partial seizures during the 4-week baseline period and at least 4 partial seizures during the 4 weeks prior to the baseline period.
* Cohort 1 patients must be receiving stable treatment with 1 or a maximum of 2 AEDs.Cohort 2 patients must be receiving stable treatment with 1, 2, or 3 AEDs.

Exclusion Criteria:

* Presence of only non-motor simple partial seizures.
* History of psychogenic seizures.
* Absences, myoclonic seizures e.g. in the context of primary generalized epilepsy.
* Previous history of Lennox-Gastaut syndrome.
* Status epilepticus or seizure clusters, according to the judgement of the investigator, occurring within 52 weeks prior to randomization.
* Pregnant or nursing (lactating) women.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To detect a dose-response by measuring the percent change in seizure frequency of BGG492 from baseline to maintenance period. | 28 days

SECONDARY OUTCOMES:
To evaluate the efficacy of BGG492 compared to placebo as a change in seizure frequency from baseline period to maintenance period. | 28 days
Responder rate: analysis of patients with a 50% or greater reduction in seizure frequency of BGG492 during the maintenance period. | 28 days
Safety and tolerability of BGG492 compared to placebo. | 12 weeks
Pharmacokinetic profile of BGG492 | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (14):
  - Barrow Neurological Clinics at St. Joseph's Hospital and MC, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Medical Center of the Rockies, Loveland, Colorado
  - AMO Corporation, Tallahassee, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Investigative Site - Private Practice, Ocean Springs, Mississippi
  - St.John's Research Institute, Inc, Springfield, Missouri
  - Renown Institute for Neurosciences, Reno, Nevada
  - NJ to Capital Health in Hamilton, Somerset, New Jersey
  - Princeton and Rutgers Neurology, Somerset, New Jersey
  - NYU Comprehensive Epilepsy Center, New York, New York
  - Thomas Jefferson University, Dept. of Psychiatry & Neurology, Philadelphia, Pennsylvania
  - Neurological Clinic of Texas, Dallas, Texas
- Novartis Investigative Site, Sofia, Bulgaria
- Germany (8):
  - Novartis Investigative Site, Bernau
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Kehl-Kork
  - Novartis Investigative Site, Marburg
  - Novartis Investigative SIte, Regensburg
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Szombathely
- Italy (6):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Catanzaro
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Venezia
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
- Slovakia (3):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- Novartis Investigative Site, Seoul, South Korea
- Switzerland (3):
  - Novartis Investigative Site, Aarau
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- Taiwan (4):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Lin-ko
  - Novartis Investigative Site, Taipei

REFERENCES:
- See also: Results for CBGG492A2207 on the Novartis clinical trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7124